CLINICAL TRIAL: NCT03435835
Title: Heat Therapy to Reduce Leg Pain and Improve Walking Tolerance in Patients With Symptomatic Peripheral Artery Disease
Brief Title: Heat Therapy to Reduce Pain and Improve Walking Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Roseguini, Bruno, PhD (Individual); Michael Emery, MD (Unknown)
Responsible Party: Principal Investigator, Raghu Motaganahalli, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1708785351
Record Dates: First submitted 2017-10-27; First posted 2018-02-19 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will not be told outright which therapy there are receiving (thermoneutral or HT) and the Cardiologist supervising the exercise test will not be told which therapy was given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham, then heat therapy (Experimental): Participants were fitted with liquid-circulating trousers. In the sham-treatment session, water at 33℃ was circulated through the trousers for 90 min using a water pump (HTP-1500, Adroit Medical, Louden, Tennessee, United States). At least 72 hrs after completion of the sham treatment session, participants returned to the laboratory and received the heat therapy (HT) treatment. In the HT session, water at 43℃ was circulated through the tube-lined trousers using a heated bath circulator (HT; Aqua Relief Systems, Akron, Ohio, United States) with the goal of increasing leg skin temperature to 37-38ºC.
  Interventions: Device: Control/Sham Treatment; Device: Heat Therapy (HT)
- Heat therapy, then sham (Experimental): Participants were fitted with liquid-circulating trousers. In the HT session, water at 43℃ was circulated through the tube-lined trousers using a heated bath circulator (HT; Aqua Relief Systems, Akron, Ohio, United States) with the goal of increasing leg skin temperature to 37-38ºC. At least 72 hrs after completion of the sham treatment session, participants returned to the laboratory and received the sham treatment. In the sham-treatment session, water at 33℃ was circulated through the trousers for 90 min using a water pump (HTP-1500, Adroit Medical, Louden, Tennessee, United States).
  Interventions: Device: Control/Sham Treatment; Device: Heat Therapy (HT)

INTERVENTIONS:
Device: Control/Sham Treatment — Water at 33ºC was circulated through water-circulating trousers.
Device: Heat Therapy (HT) — Water at 42-43ºC was circulated through the water-circulating trousers.

SUMMARY:
The purpose of this study is to investigate whether exposure to heat therapy improves calf muscle oxygenation and enhances walking tolerance in patients with symptomatic Peripheral Arterial Disease (PAD).

DETAILED DESCRIPTION:
Heat therapy (HT) is an emerging non-invasive approach that has been shown to enhance vascular function of the leg in old individuals. The objective of this study is to establish evidence to support the validity of HT in improving walking tolerance on PAD patents.

Subjects will complete baseline assessments for eligibility, including medical history and ankle-brachial measurement. Eligible participants will be asked to report to the laboratory on 4 different occasions. The purpose of visits 1 and 2 The central hypothesis of this study, based on preliminary data, is that exposure to HT will enhance the oxygenation of calf muscles during exercise and as a result, the onset of pain will be delayed and walking performance will be enhanced. is to familiarize the participants with the treadmill walking test and assess the test-retest reliability of maximal walking time determination. On visits 3 and 4 participants will receive either heat treatment or a control treatment for 80 min prior to undergoing a symptom-limited incremental test on the treadmill.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with stable symptomatic leg claudication for 6 months or longer.
* Ankle brachial index < 0.9

Exclusion Criteria:

* Heart Failure
* COPD
* Critical limb ischemia
* Prior amputation
* Exercise-limiting co-morbidity
* Recent infrainguinal revascularization or planned during study period
* Plans to change medical therapy during duration of the study
* Active cancer
* Chronic kidney disease
* HIV positive, active HBV or HCV disease
* Presence of any unsuitable comorbid clinical condition in the opinion of the PI
* Peripheral neuropathy, numbness or paresthesia in the legs
* Morbid obesity, BMI > 36 or unable to fit in water-circulating pants
* Open wounds or ulcers on the extremity
* Unable to walk on the treadmill

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raghu L Motaganahalli, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified and contacted by the Indiana Clinical and Translational Science Institute Research Network (ResNet) research assistants. After interest in participation was established, patients were contacted directly by the investigators. Additional study participants were identified by physicians from the Division of Vascular Surgery at Methodist Hospital.
Pre-assignment Details: Nineteen participants were consented, but three were withdrawn before receiving an experimental treatment due to the inability to safely and consistently perform the treadmill exercise test. A total of 16 participants completed all study visits.
Groups:
- Sham, Then Heat Therapy: Participants were fitted with liquid-circulating trousers. In the sham treatment session, water at 33℃ was circulated through the trousers for 90 min using a water pump (HTP-1500, Adroit Medical, Louden, Tennessee, United States). At least 72 hrs following the completion of the sham treatment, patients returned to the laboratory and underwent the leg heat therapy (HT treatment). In the HT session, water at 43℃ was circulated through the tube-lined trousers using a heated bath circulator (HT; Aqua Relief Systems, Akron, Ohio, United States) with the goal of increasing leg skin temperature to 37-38ºC.
- Heat Therapy, Then Sham: Participants were fitted with liquid-circulating trousers. In the HT session, water at 43℃ was circulated through the tube-lined trousers using a heated bath circulator (HT; Aqua Relief Systems, Akron, Ohio, United States) with the goal of increasing leg skin temperature to 37-38ºC. At least 72 hrs following the completion of the HT treatment, patients returned to the laboratory and underwent the sham treatment. In the sham treatment session, water at 33℃ was circulated through the trousers for 90 min using a water pump (HTP-1500, Adroit Medical, Louden, Tennessee, United States).
Period: First Intervention
Arm/Group | Sham, Then Heat Therapy | Heat Therapy, Then Sham
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout
Arm/Group | Sham, Then Heat Therapy | Heat Therapy, Then Sham
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Sham, Then Heat Therapy | Heat Therapy, Then Sham
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Nineteen participants were consented, but three were withdrawn before receiving an experimental treatment due to inability to safely and consistently perform the treadmill exercise test. Baseline clinical characteristics of the 16 participants that completed all study visits are presented.
Groups:
- All Study Participants: Participants were assigned, using a randomized, crossover design, to undergo a single session of either a sham treatment (sham) or heat therapy (HT) prior to a symptom-limited cardiopulmonary treadmill exercise test. In the sham treatment session, water at 33°C was circulated through the trousers for 90 min using a water pump (HTP-1500, Adroit Medical, Louden, Tennessee, United States). In the HT session, water at 43℃ was circulated through the tube-lined trousers using a heated bath circulator (HT; Aqua Relief Systems, Akron, Ohio, United States) with the goal of increasing leg skin temperature to 37-38ºC.
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Peak Walking Time
Description: Exercise testing was performed in a motorized treadmill (Pro 27, Woodway, St. Paul, Minnesota, United States) following the Gardner-Skinner protocol, which consists of walking at a constant speed (2 mph) with a 2%-grade increase every 2 min (Gardner et al., 1991). Participants received standardized instructions and were asked to indicate when they first began to feel leg pain with a "thumbs up" signal (defined as COT), and then give a "thumbs down" signal when they could no longer continue with the test (defined as PWT).
Time Frame: Immediately after exposure to a single session of heat therapy or sham treatment, up to ~20 min
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Sham Treatment: Participants were fitted with liquid-circulating trousers and water at 33°C was circulated through the trousers for 90 min using a water pump (HTP-1500, Adroit Medical, Louden, Tennessee, United States).
- Heat Therapy: Participants were fitted with liquid-circulating trousers and water at 43°C was circulated through the tube-lined trousers for 90 min using a heated bath circulator (HT; Aqua Relief Systems, Akron, Ohio, United States) with the goal of increasing leg skin temperature to 37°C-38°C.
Arm/Group | Sham Treatment | Heat Therapy
Number analyzed (Participants) | 16 | 16
seconds | 955.6 (84.3) | 947.7 (88.1)

2. Secondary Outcome: Claudication Onset Time
Description: as for outcome 1
Time Frame: The exercise test was performed immediately after exposure to a single session of either heat therapy or sham, up to ~20 min
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Sham Treatment | Heat Therapy
Number analyzed (Participants) | 16 | 16
Seconds | 452.6 (53.2) | 442.9 (65.1)

3. Secondary Outcome: Peak Systolic Blood Pressure
Description: Blood pressure was measured in the left arm using a stethoscope and sphygmomanometer during exercise.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Treatment | Heat Therapy
Number analyzed (Participants) | 16 | 16
mmHg | 193.3 (23.2) | 189.3 (31.0)

4. Secondary Outcome: Peak Diastolic Blood Pressure
Description: Blood pressure was measured in the left arm using a stethoscope and sphygmomanometer prior and during exercise
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham Treatment | Heat Therapy
Number analyzed (Participants) | 16 | 16
mmHg | 74.2 (9.7) | 73.5 (11.6)

5. Secondary Outcome: Peak Calf Tissue Saturation Index
Description: The tissue saturation index (TSI%) of the most symptomatic leg was assessed with a commercially available NIRS system (Portamon, Artinis Medical Systems, The Netherlands).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: % tissue saturation
Arm/Group | Sham Treatment | Heat Therapy
Number analyzed (Participants) | 14 | 14
% tissue saturation | 43.9 (7.6) | 43.1 (8.2)

6. Secondary Outcome: Post-exercise Plasma Endothelin-1 Concentration
Description: Commercially available enzyme-linked immunosorbent assay kits were used to measure the plasma concentrations of ET-1 (DET100, Endothelin-1 Quantikine ELISA Kit, R&D Systems, Minneapolis, MN, United States)
Time Frame: The exercise test was performed immediately after exposure to a single session of either heat therapy or sham, up to ~20 min. Ten minutes following completion of the incremental treadmill test, blood samples were obtained for the assessment of serum ET-1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sham Treatment | Heat Therapy
Number analyzed (Participants) | 14 | 14
pg/mL | 2.0 (0.6) | 1.7 (0.5)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study (approximately 1 month).
Arm/Group | Sham Treatment | Heat Therapy
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Treatment (N=16) | Heat Therapy (N=16)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 0 — Baseline blood draw indicated that participant had plasma potassium concentration of 2.9 (critical value). The study session was stopped and the patient was escorted to the Emergency Department.
Hypotension (Vascular disorders) | 0 | 1 — After the third blood draw the patient became lightheaded, the blood pressure was 86/50.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT03435835/Prot_SAP_000.pdf